CLINICAL TRIAL: NCT04435275
Title: Development of an Automated and Scalable Virtual Assistant to Aid in PPE Adherence and Clinical Protocols for Healthcare Worker Safety
Brief Title: Virtual Assistant for COVID-19 PPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-5399
Record Dates: First submitted 2020-06-09; First posted 2020-06-17 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: PPE adherence
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Donning PPE using VA then doffing PPE using HC (Active Comparator): Study subjects will receive VA guidance for donning first, then guidance from a human coach (HC) for doffing.
  Interventions: Other: Virtual Assistant first, then Human Coach
- Donning PPE using HC then doffing PPE using VA (Active Comparator): Study subjects will receive HC guidance for donning first, then VA guidance for doffing.
  Interventions: Other: Human Coach first, then Virtual Assistant
- Intubation using VA then extubation using HC; (Active Comparator): Study subjects will receive VA guidance for the intubation first , then HC guidance for extubation procedure
  Interventions: Other: Virtual Assistant first, then Human Coach
- Intubation using HC then extubation using VA (Active Comparator): Study subjects will receive HC guidance for the intubation first , then VA guidance for extubation procedure
  Interventions: Other: Human Coach first, then Virtual Assistant

INTERVENTIONS:
Other: Virtual Assistant first, then Human Coach — Instructions to aid healthcare worker adherence to proper PPE and intubation and extubation procedure is given by a VA (e-coach) in place of a safety officer (a human coach).
  Arms: Donning PPE using VA then doffing PPE using HC; Intubation using VA then extubation using HC;
Other: Human Coach first, then Virtual Assistant — instructions to aid healthcare worker adherence to proper PPE and intubation and extubation procedure is given by a safety officer (a human coach).
  Arms: Donning PPE using HC then doffing PPE using VA; Intubation using HC then extubation using VA

SUMMARY:
The COVID virus is acquired through droplet and micro droplet transmission. Although healthcare workers must adhere to strict up-to-date clinical procedures to minimize exposure to the virus and avoid contamination, the assumption that everyone can precisely remember every step is improbable as many of these procedures are quite complex and involve multiple steps in stressful situations. Further the use of a trained safety officer to ensure adherence is not always feasible due to the ever growing demand of healthcare providers. Investigators propose to utilize the Amazon Alexa device and Alexa Skills application to develop a voice enabled virtual assistant to guide healthcare professionals through the exact steps of clinical procedures including the donning and doffing of PPE, intubation and extubation procedures.

Methods A total of 10 staff anesthesiologists will be recruited to participate in phase 1 of the study to evaluate the utility and functionality of this VA device.

A total of 40 healthcare professionals will be recruited to participate in phase 2 of the study. Anesthesia providers (staff and fellows), anesthesia assistants, respiratory assistants and operating room nurses will be randomized to receive instructional guidance by the VA on one test occasion and a human coach on another occasion. During this phase of the study, the effectiveness of this VA prototype will be compared with a trained human safety officer / coach in its ability to provide instructional guidance for 4 safety and clinical procedures: 1) proper donning of personal protective equipment (PPE); 2) doffing of PPE; 3) intubation (putting in a breathing tube) and 4) extubation (taking out a breathing tube).

ELIGIBILITY:
Inclusion Criteria:

* Only anesthesia attending staff are allowed in the phase 1 study.
* Any working anesthesia staff and fellow, anesthesia assistant, respiratory assistant and operating room nurse are qualified to take part in phase 2 of this study. However, only anesthesia staff and fellows and anesthesia assistants will participate in the part that involves intubation and extubation.

Exclusion Criteria:

• Unwillingness to enter the study for phase 1 or phase 2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
performance of healthcare workers | 0- 30mins during donning
  Errors occurred during donning of PPE measured by procedure checklist
performance of healthcare workers | 0- 30mins during doffing
  Errors occurred during doffing of PPE measured by procedure checklist
performance of healthcare workers | 0- 30mins during intubation
  Errors occurred during intubation measured by procedure checklist
performance of healthcare workers | 0- 30mins during extubation
  Errors occurred during extubation measured by procedure checklist

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada